CLINICAL TRIAL: NCT00721032
Title: Anti-arrhythmic Medication v. MRI-Merge Ablation in the Treatment of Ventricular Tachycardia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00011012
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular tachycardia (VT); Implantable cardioverter-defibrillator (ICD); Ablation; Cardiomyopathy; Electrophysiology study
MeSH Terms: conditions — Tachycardia, Ventricular; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Magnetic resonance imaging (MRI)-guided ablation of ventricular tachycardia.
  Interventions: Procedure: MRI guided VT ablation
- 2 (Active Comparator): Anti-arrhythmic group.
  Interventions: Drug: Increased dose of amiodarone

INTERVENTIONS:
Procedure: MRI guided VT ablation — Magnetic resonance imaging (MRI)-guided ablation of ventricular tachycardia (VT)
  Arms: 1
Drug: Increased dose of amiodarone — Increase the dose of amiodarone according to the following scheme:
  current dose -> new dose 100 once daily (QD) -> 200 QD; 200 QD -> 400 QD; 300 QD -> 600 QD; 400 QD -> 600 QD
  Arms: 2

SUMMARY:
Ventricular tachycardia (VT) is a morbid arrhythmia responsible for many sudden deaths and ICD shocks. Despite much progress in the treatment of arrhythmia, VT remains a therapeutic challenge. Most patients with VT have an implantable cardioverter defibrillator (ICD) for secondary prevention of sudden cardiac death, however, an ICD merely treats VT, it does not prevent VT. In patients with recurrent VT and ICD shocks, two strategies are available to decrease the burden of VT. The first is antiarrhythmic drugs, and the second is VT ablation. The aim of this study is to compare the efficacy of antiarrhythmic drugs and VT ablation guided by MRI. VT can sometimes be suppressed with antiarrhythmic medications, however, these are often ineffective, and carry a high burden of side effects. Many forms of VT can be cured by selective destruction of critical electrical pathways with catheter ablation. A major limitation in the ablation of VT, however, is the time required to localize scar tissue and important pathways for targeting of lesions. Magnetic resonance imaging can now obtain reliable images of scar location within the ventricles. Recent advances in electroanatomical mapping systems allow operators to import pre-acquired images into the mapping system. The aim of this study is to examine the feasibility of importing historic MRI scar maps of the ventricles into the electroanatomical system and using such images to guide catheter ablation, as compared to antiarrhythmic drug suppression of VT. We suspect that MRI guidance will be especially useful in patients with "unstable" VT, i.e. VT that causes an abrupt drop in blood pressure, and thus cannot be maintained in the electrophysiology (EP) lab for mapping and entertainment purposes. Patients referred for VT ablation have ICDs. Through previously completed animal work (Circulation 2004; 110(5): 475-82) and a human trial (2006 Sep 19;114(12):1277-84) we have demonstrated the safety of MRI in the setting of pacemakers and implantable defibrillators using appropriate precautions. Through careful device programming and using MRI sequences with limited energy exposure (specific absorption rate < 2 W/kg) we will study the pre procedural myocardial anatomy of patients enrolled into this study.

The primary endpoint will be lack of VT documented by implantable defibrillator (when present) interrogation or Holter monitoring 6 months post ablation. The secondary endpoints will be comparison of inducible arrhythmia at the end of the procedure, procedure time, comparison of endocardial voltage mapping to scar on delayed enhancement MRI images, and complications in each study arm.

ELIGIBILITY:
Inclusion:

* Current treatment with amiodarone
* Ischemic or non-ischemic cardiomyopathy
* Monomorphic ventricular tachycardia at any cycle length, with > 1 occurrence of the same cycle length and morphology, at least one episode needs to be of sufficient duration to result in a shock.
* No contraindication to up titration of meds or to VT radiofrequency ablation (RFA)

Exclusion:

* Primary antiarrhythmic medication other than amiodarone
* Amiodarone at dose of 600 mg daily or higher
* Polymorphic VT as culprit rhythm
* History of metal exposure (welding)
* Pregnant women
* Recent myocardial infarction
* Planned coronary revascularization
* Implantable cardiac devices not previously tested for safety in the setting of MRI
* Glomerular Filtration Rate (GFR) < 30 ml/min

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Freedom from ventricular tachycardia documented by implantable defibrillator cardioverter 6 months post ablation. | 6 months

SECONDARY OUTCOMES:
inducible arrhythmia at the end of the procedure, | During procedure
Procedure time | During procedure
Comparison of endocardial voltage mapping to scar on delayed enhancement MRI images | During procedure
Complications of the procedure | 30 days following procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States